CLINICAL TRIAL: NCT00947219
Title: A Randomized, Double-Blind, Control Device Clinical Trial to Evaluate the Safety and Efficacy of the HairMax LaserComb 2009, 9 & 12 Beam Models: For the Treatment of Androgenetic Alopecia in Males
Brief Title: Treatment of Androgenic Alopecia in Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9.12 2009-M-02
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Androgenetic Alopecia; Hair Loss; Male Pattern Baldness
Keywords: Androgenetic Alopecia; Hair Loss; Male Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HairMax LaserComb 2009, 12 Beam (Active Comparator): Low Level Laser Medical Device 2009 with 12 laser beams
  Interventions: Device: HairMax LaserComb
- HairMax LaserComb 2009 9 Beam (Active Comparator): Low Level Laser Mecial Device 2009 with 9 laser beams
  Interventions: Device: HairMax LaserComb
- Control device (Active Comparator): The control device appears identical to the active device, but utilizes 9 LED lights instead of laser lights. The randomized devices are blinded to the study investigator and distributed in a blinded manner to the participants.
  Interventions: Device: Control device

INTERVENTIONS:
Device: HairMax LaserComb — Device application 3 times week (non-consecutive days), for 26 weeks
  Arms: HairMax LaserComb 2009 9 Beam; HairMax LaserComb 2009, 12 Beam
Device: Control device — Device is used 3 times a week on non-consecutive days
  Arms: Control device

SUMMARY:
The purpose of this study is to evaluate the change in terminal hair count at 16 and 26 weeks compared to baseline measurements.

DETAILED DESCRIPTION:
This is randomized, double-blind, control device clinical study across 3 sites, evaluating changes in terminal hair-count in the evaluation zone having evidence of androgenetic alopecia (miniaturized hair).

The trial will involve approximately 75 male subjects who have been diagnosed with androgenetic alopecia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types I-IV, with classifications of Norwood-Hamilton IIa to V, have active hair loss within the last 12 months.

Subjects will use the device on three non-consecutive days a week as directed per device for 26 weeks treatment duration.

Safety analysis will be assessed based on the reports of adverse events during study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of androgenetic alopecia
* Fitzpatrick Skin Types I-IV
* Norwood-Hamilton IIa to V
* Active hair loss within last 12 months

Exclusion Criteria:

* Photosensitivity to laser light
* Malignancy in the target area

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Draelos, MD, Principal Investigator — High Point, NC; David Goldberg, M.D., Principal Investigator — Skin & Laser; Abe Marcadis, M.D., Principal Investigator — Palm Beach Research
Locations (3):
- United States (3):
  - Abe Marcadis, M.D., West Palm Beach, Florida
  - David Goldberg, M.D., Hackensack, New Jersey
  - Zoe Draelos, M.D., High Point, North Carolina

REFERENCES:
- [Background] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male subjects who have been diagnosed with androgenetic alopicia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types i-IV and Norwood Hamilton Classifications of IIa to IV and have active hair loss with the last 12 months
Pre-assignment Details: Exclusion criteria: Individuals with photosensitivity to laser light, history of any malignancy in target area, has used phytotherapy (e.g. saw palmetto) with 8 weeks prior to baseline. Subjects who has chronic dermatological conditions (eczema, psoriasis, etc) of the scalp other than male pattern baldness
Groups:
- HairMax LaserComb 2009, 12 Beam: LLLT Device 2009 12 Beam, Control Device
- HairMax LaserComb 2009 9 Beam: LLLT Device 2009 9 Beam, Control Device
- Control Device: Control device emitting LED light
Period: Overall Study
Arm/Group | HairMax LaserComb 2009, 12 Beam | HairMax LaserComb 2009 9 Beam | Control Device
Started | 28 | 25 | 26
Completed | 22 | 21 | 22
Not Completed | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HairMax LaserComb 2009, 12 Beam | HairMax LaserComb 2009 9 Beam | Control Device | Total
Number analyzed (Participants) | 28 | 25 | 26 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 26 | 79
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 28 | 25 | 26 | 79

OUTCOME MEASURES:

1. Primary Outcome: Changes in Terminal Hair Count at 16 and 26 Weeks Compared to Baseline in Men Diagnosed With Androgenetic Alopecia
Description: The primary analysis of effectiveness was an analysis of covariance, which separately modeled terminal hair count at Week 16 and Week 26 as a function of treatment group (HairMax LaserComb 2009 9 Beam vs.control), study center, age (as a continuous variable), and Fitzpatrick Skin Type classification (as a categorical variable with four levels). The active group was compared to the control device using least squares means with a two-sided test at the 5% level of significance.
Time Frame: baseline, 16 and 26 weeks
Measure: Mean (Standard Deviation); unit: hairs per cm^2
Units Other Than Participants: hairs per cm^2
Groups:
- HairMax LaserComb 2009, 12 Beam: The active LLLT Device 2009 with 12 laser modules
- HairMax LaserComb 2009 9 Beam: the active LLLT Device 2009 9 laser modules
- Control Device: Control device emitting white light
Arm/Group | HairMax LaserComb 2009, 12 Beam | HairMax LaserComb 2009 9 Beam | Control Device
Number analyzed (Participants) | 22 | 21 | 22
Number analyzed (hairs per cm^2) | 22 | 21 | 22
hairs per cm^2
  Change at 16 weeks | 23.5 (17.67) | 20.4 (14.52) | 4.4 (8.38)
  Change at 26 weeks | 25.7 (16.92) | 20.9 (14.08) | 9.4 (12.94)

ADVERSE EVENTS:
Arm/Group | HairMax LaserComb 2009, 12 Beam | HairMax LaserComb 2009 9 Beam | Control Device
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No